CLINICAL TRIAL: NCT00001874
Title: Technical Evaluation of Cardiovascular Magnetic Resonance Imaging and Spectroscopy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990048; 99-H-0048
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-03

CONDITIONS: Cardiovascular Disease; Healthy
Keywords: Imaging; Spectroscopy; MRI; Cardiovascular; Technical Development; Safety; Gadolinium; Heart; Toxicity; Adverse Events; Normal Volunteer
MeSH Terms: conditions — Cardiovascular Diseases

SUMMARY:
Magnetic resonance imaging (MRI) and spectroscopy are diagnostic tools that create high quality images of the human body without the use of X-ray (radiation). MRI uses different levels of magnetic fields to create images of the body and organs. Occasionally, researchers will give patients undergoing a MRI an injection of a contrast substance. The contrast substance works by brightening areas of the magnetic resonance image.

In this study researchers plan to use magnetic resonance imaging with contrast substances and exercise on normal volunteers in order to evaluate different aspects of its performance. Information gathered from this study may be used to develop more specific research studies involving MRI....

DETAILED DESCRIPTION:
Technical evaluation of magnetic resonance imaging and spectroscopy will be performed on normal volunteers. These studies will be conducted in the NIH MRI systems located in Suburban Hospital in Bethesda, Maryland. These studies may involve the intravenous administration of commercially available MR contrast media and exercise. The results will be used to evaluate the performance of various pulse sequences, gradient coils, and RF coils on human subjects and will provide essential ground work for specific patient protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any normal volunteer above the age 18 who is capable of giving informed consent will be included.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contradiction to MR scanning.

1. Brain aneurysm clip
2. Implanted neural stimulator
3. Implanted cardiac pacemaker implanted defibrillator
4. Cochlear implant
5. Ocular foreign body (e.g. metal shavings)
6. Insulin pump
7. Pregnant women (when uncertain, subjects will undergo urine or blood testing).
8. Kidney
9. Paralyzed hemidiaphragm
10. Morbid obesity
11. Claustrophobia
12. Any condition in the PI's judgement which present unncessary risk

EXCLUSION CRITERIA FOR GADOLINIUM ENHANCED STUDIES:

1. Lactating women
2. Subjects with hemoglobinopathies
3. Asthma
4. Renal or hepatic disease

Subjects will be excluded if it is deemed that they have a condition that would preclude their use for technical development (e.g. paralyzed hemidiaphragm, morbid obesity, claustrophobia etc.) or present unnecessary risk (e.g. pregnancy, surgery of uncertain type, etc.).

Lactating women and subjects with hemoglobinopathies, asthma, or renal or hepatic disease will be excluded from studies involving the adminstration of contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1999-02-22; Primary Completion 2009-08-03 (Actual); Study Completion 2009-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

REFERENCES:
- [Background] Frank JA, Mattay VS, Duyn J, Sobering G, Barrios FA, Zigun J, Sexton R, Kwok P, Woo J, Moonen C, et al. Measurement of relative cerebral blood volume changes with visual stimulation by 'double-dose' gadopentetate-dimeglumine-enhanced dynamic magnetic resonance imaging. Invest Radiol. 1994 Jun;29 Suppl 2:S157-60. doi: 10.1097/00004424-199406001-00052. No abstract available. PMID 7928216
- [Background] Mattay VS, Weinberger DR, Barrios FA, Sobering GS, Kotrla KJ, van Gelderen P, Duyn JH, Sexton RH, Moonen CT, Frank JA. Brain mapping with functional MR imaging: comparison of gradient-echo--based exogenous and endogenous contrast techniques. Radiology. 1995 Mar;194(3):687-91. doi: 10.1148/radiology.194.3.7862963.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423